CLINICAL TRIAL: NCT00180921
Title: Phase II Study of Imatinib (Glivec) Administered as a Daily Oral Treatment in Patients With Recurrent/Metastatic Adenoid Cystic Carcinoma of the Head and Neck Overexpressing KIT
Brief Title: Study of Imatinib (Glivec) in Patients With Adenoid Cystic Carcinoma of the Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI BFR 17
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2006-09

CONDITIONS: Cancer of the Head and Neck; Carcinoma, Adenoid Cystic
Keywords: Adenoid cystic carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Adenoid Cystic | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib

SUMMARY:
This is a Phase II study of imatinib (Glivec) administered as a daily oral treatment in patients with recurrent/metastatic adenoid cystic carcinoma of the head and neck overexpressing KIT.

DETAILED DESCRIPTION:
Patients with relapsing and/or metastatic adenoid cystic carcinoma of the salivary gland of the head and neck are usually poor responders to conventional cytotoxic chemotherapy.

The investigation of proliferation pathways involving tyrosine kinase receptors such as c-kit receptor (KIT) and PDGF receptor may allow to identify a molecular target for novel therapeutic approaches in patients with adenoid cystic carcinoma who failed locoregional treatment.

Several publications in the literature and the pathological study we conducted in Institut Gustave Roussy show that KIT overexpression is observed in at least 80-90% of the cases of adenoid cystic carcinoma, supporting the investigation of imatinib in patients with adenoid cystic carcinoma overexpressing KIT.

Imatinib is an orally administrated, well tolerated compound that could be given on an outpatient schedule to patients with relapsing/metastatic adenoid cystic carcinoma of the head and neck.

Because of the infrequent occurrence of salivary gland malignancies, a multicenter trial will be mandatory and the study will include at least 2 centers represented by Institut Gustave Roussy, Villejuif; and Hôpital Georges-Pompidou, Paris.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenoid cystic carcinoma overexpressing KIT (by immunohistochemistry) with recurrent disease documented by computed tomography (CT) scan or magnetic resonance imaging (MRI).
* Presence of at least one dimensionally measurable target lesion (contrast enhancing lesion with the largest diameter >= 2 cm, based on CT or MRI scan done within 4 weeks before the start of treatment).
* Patients able to swallow an oral compound.
* World Health Organization (WHO) performance status < 2.
* Life expectancy of >= 3 months.
* Aged >= 18 years.
* Normal hematological (neutrophils >= 1.5 x 10^9 cells/l, platelets >= 100 x 10^9 cells/l), hepatic (bilirubin < 1.5 times the upper limit of the normal range; alkaline phosphatase and transaminases <= 2.5 x the upper limit of the normal range) and renal (serum creatinine <= 150 mmol/l) functions.
* Written informed consent.

Exclusion Criteria:

* Abnormal cardiac function with history of ischaemic heart disease in the past 6 months and/or abnormal 12 lead electrocardiogram (ECG).
* Previous or current malignancies at other sites with the exception of cone biopsied carcinoma of the cervix and adequately treated basal or squamous cell skin carcinoma.
* Concomitant treatment with warfarin or any other anticoagulants.
* Unstable systemic diseases or active uncontrolled infections.
* Patients (male and female) not using effective contraception if of reproductive potential.
* Females pregnant or lactating or positive beta human chorionic gonadotropin (bHCG) at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-07

PRIMARY OUTCOMES:
To assess progression-free survival under treatment with imatinib mesylate in patients with relapsing/metastatic adenoid cystic carcinoma of the head and neck overexpressing KIT. | at 6 months

SECONDARY OUTCOMES:
The secondary objectives are to estimate the objective response rate (Response Evaluation Criteria in Solid Tumors [RECIST] criteria), disease control and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Faivre, MD, Principal Investigator — Centre Hospitalier de Beaujon
Locations (1):
- Institut Gustave Roussy, Villejuif, France